CLINICAL TRIAL: NCT05907343
Title: Closed-Loop Brain Stimulation as a Potential Intervention for Cognitive Decline
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Jose del R. Millan, Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00003055
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Mild Cognitive Impairment
Keywords: MCI; Older adults; Cognitive control; Memory impairment
MeSH Terms: conditions — Cognitive Dysfunction; Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Sham TBS (Active Comparator)
  Interventions: Device: Sham TBS
- Closed-Loop TBS (Active Comparator)
  Interventions: Device: Closed-loop TBS
- Open-Loop TBS (Active Comparator)
  Interventions: Device: Open-loop TBS

INTERVENTIONS:
Device: Sham TBS — A BCI records and analyzes the participant's EEG as they perform cognitively demanding video game tasks. The BCI delivers TBS with a sham coil when its output indicates that the participant is not properly engaged in the video game.
  Arms: Sham TBS
Device: Closed-loop TBS — A BCI records and analyzes the participant's EEG as they perform cognitively demanding video game tasks. The BCI delivers TBS with a real coil when its output indicates that the participant is not properly engaged in the video game.
  Arms: Closed-Loop TBS
Device: Open-loop TBS — A BCI records and analyzes the participant's EEG as they perform cognitively demanding video game tasks. TBS with the real coil is delivered irrelevant of the BCI decoder output.
  Arms: Open-Loop TBS

SUMMARY:
The goal of this clinical study is to investigate the effectiveness of non-invasive stimulation to enhance cognitive control abilities in cognitively healthy adults and older adults diagnosed with mild cognitive disorder (MCI). The main questions it aims to answer are:

* whether it is possible to restore various cognitive functions in older adults diagnosed with MCI by delivering theta burst stimulation (TBS), a form of transcranial magnetic stimulation, and
* whether closed-loop TBS is able to induce therapeutic benefits that outperform open-loop TBS.

Participants play a cognitive video game while a brain-computer interface (BCI) analyzes their electroencephalogram (EEG) signals and decodes the presence or absence of the contingent negative variation (CNV) potential, a marker of cognitive control. The BCI triggers TBS when its outputs indicate that the participant is not engaged properly in the video game.

Researchers will compare the effects of sham, closed-loop, and open-loop TBS using the outcome metrics described below to see how much cognitive restorations is achievable with each stimulation modality.

ELIGIBILITY:
Inclusion Criteria:

* Cognitively normal younger adults

  1. Ages between 18 to 35 years
  2. Good general health
  3. Normal or corrected vision
  4. Completed elementary school education or able to understand middle school level experiment instructions
* Cognitively normal older adults

  1. Ages between 60 to 90 years
  2. Good general health
  3. Normal or corrected vision
  4. Completed elementary school education or able to understand middle school level experiment instructions
  5. Score of 23 or higher on the Montreal Cognitive Assessment, a brief formal cognitive screening test, which is used to indicate absence of cognitive impairment
* Older adults with mild cognitive impairment (MCI)

  1. Ages between 60 to 90 years
  2. Diagnosis of MCI according to the National Institute on Aging - Alzheimer's Association (NIA-AA) criteria
  3. Good general health
  4. Normal or corrected vision
  5. Completed elementary school education or able to understand middle school level experiment instructions

Exclusion Criteria:

1. Neurological or psychiatric diseases (e.g., personal history of epilepsy/seizure brain damage, multiple sclerosis, schizophrenia, substance use disorder, etc.).
2. Current use of psychotropic medications with cognitive side effects (e.g., benzodiazepines, anticonvulsants, antipsychotics, etc.)
3. Current use of cognitive enhancing medications (e.g., Adderall, Memantine, etc.)
4. Factors hindering EEG acquisition and TMS delivery (e.g., skin infection, wounds, dermatitis, etc.)
5. Factors hindering MRI acquisition (e.g., implants, metallic tattoos, etc.)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Behavioral performance of the video game task | Up to 1 hour after intervention
  The behavioral performance, pressing or not pressing a button, reflects the level of cognitive control performance of the subjects. It measures whether the participants made a correct decision, and their response time, in a given trial.
Accuracy of the BCI classifier output | Up to 1 hour after intervention
  The BCI classifier output reflects the presence or absence of the cognitive EEG patterns elicited during the cognitive videogame tasks. For each participant, the BCI outputs will be compared to their behavioral responses (pressing or not pressing a button).
Cognitive assessment I: Montreal Cognitive Assessment | Up to 8 weeks after intervention
  Telephone version, Score range: 0 - 22* (Units on a Scale)
  (* high scores = better)
Cognitive assessment II: Hopkins Adult Reading Test | Up to 8 weeks after intervention
  Score range: 70 - 131* (Units on a Scale)
  (* high scores = better)
Cognitive assessment III: Multilingual Naming Test | Up to 8 weeks after intervention
  Score range: 0 - 32* (Units on a Scale)
  (* high scores = better)
Cognitive assessment IV: Animal Naming | Up to 8 weeks after intervention
  Score range: 0 - 40* (Units on a Scale)
  (* high scores = better)
Cognitive assessment V: Number Span | Up to 8 weeks after intervention
  * Forward, Score range: 0 - 14* (Units on a Scale)
  * Backward, Score range: 0 - 14* (Units on a Scale)
  (* high scores = better)
Cognitive assessment VI: Trail Making Test | Up to 8 weeks after intervention
  Parts A and B, Score range: 10 - 300** (Units on a Scale)
  (** high scores = worse)
Cognitive assessment VII: Southwestern Assessment of Processing Speed | Up to 8 weeks after intervention
  Score range: 0 - 75* (Units on a Scale)
  (* high scores = better)
Cognitive assessment VIII: Hopkins Verbal Learning Test-Revised | Up to 8 weeks after intervention
  * Immediate Total, Score range: 0 - 36* (Units on a Scale)
  * Delayed Recall, Score range:0 - 12* (Units on a Scale)
  * Percent Retention, Score range:0 - 100* (Units on a Scale)
  (* high scores = better)
Cognitive assessment IX: Brief Visuospatial Memory Test-Revised | Up to 8 weeks after intervention
  * Immediate Total, Score range: 0 - 36* (Units on a Scale)
  * Delayed Recall, Score range:0 - 12* (Units on a Scale)
  * Percent Retention, Score range:0 - 100* (Units on a Scale)
  (* high scores = better)
Cognitive assessment X: Controlled Oral Word Association Test | Up to 8 weeks after intervention
  Score range: 0 - 80* (Units on a Scale)
  (* high scores = better)
Cognitive assessment XI: Stroop Color and Word Test | Up to 8 weeks after intervention
  * Word, Score range: 0 - 140* (Units on a Scale)
  * Color, Score range:0 - 120* (Units on a Scale)
  * Color-Word, Score range:0 - 80* (Units on a Scale)
  (* high scores = better)

CONTACTS AND LOCATIONS:
Overall Officials: José del R. Millán, PhD, Principal Investigator — University of Texas at Austin; Robin Hilsabeck, PhD, ABPP, Principal Investigator — University of Texas at Austin
Locations (1):
- Health Discovery Building, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All anonymized data will be made available by the online publication date. These data will be placed in public servers for any interested researcher to access it.
Time Frame: Data will become permanently available by the online publication date.
Access Criteria: Any interested researcher will have access.